CLINICAL TRIAL: NCT06521788
Title: Application Research of B-ultrasound Assisted by Artificial Intelligence in Breast Cancer Screening
Brief Title: Artificial Intelligence Assisted Breast Ultrasound in Breast Cancer Screening
Acronym: AIBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ying Zheng, Director of Cancer Prevention Department, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20210712
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Screening
Keywords: Cancer epidemiology; Artificial intelligence; Ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI assisted B-ultrasound breast cancer screening (Experimental): Participants aged 35-70 years will be screened for breast cancer with AI assisted B-ultrasound
  Interventions: Device: AI-assisted breast ultrasound
- routine screening (Active Comparator): Participants aged 35-70 years will be screened for breast cancer with routine B-ultrasound by experienced primary care physicians.
  Interventions: Device: Routine breast ultrasound

INTERVENTIONS:
Device: AI-assisted breast ultrasound — AI-assisted breast ultrasound in community-based breast cancer screening
  Arms: AI assisted B-ultrasound breast cancer screening
Device: Routine breast ultrasound — Routine breast ultrasound conducted by primary care physicians
  Arms: routine screening

SUMMARY:
AIBU is a randomized, open-label study assessing the effectiveness of an articificial intelligence-assisted breast ultrasound breast cancer screening strategy compared to standard screening (according to the current local guidelines in each participating area) in detecting late-stage breast cancers.

DETAILED DESCRIPTION:
we enrolled asymptomatic women Women From January 2021 to December 2022, and then followed up for the next 1 year. The main study endpoint will be measured at the end of the one year after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 35-70 who participated in breast cancer screening (Shanghai Rural Women "Women two cancer screening project", national major public health service project "Rural women breast cancer screening Project" and "Gynecological diseases and breast diseases screening project for retired and living difficult women") in Shanghai district

Exclusion Criteria:

* 1. Personal history of breast carcinoma, either invasive or ductal carcinoma in situ (DCIS); 2. Personal history of any types of malignant neoplasms; 3. Known condition or suspicion of severe cardiopulmonary insufficiency, liver and kidney insufficiency and other systemic diseases; 4. Known condition or suspicion of serious comorbidities and average life expectancy less than 5 years; 5. History of lateral or bilateral mastectomy; 6. Disagree to participate in the study and follow-up interviews.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21790 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of early breast cancer in each arm | 4 years
  Early cancers should meet any of the following criteria at the time of diagnosis: less than 20 milimeters in diameter, no metastatic lymph nodes in the axilla, no distant metastasis, non-invasive cancers, stage 0, stage I, and stage IIa IIb (T2N1M0) breast cancer according to American Joint Committee on Cancer (AJCC) 8th staging.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value of the screening methods | 4 years
  A true-positive screening result (sensitivity) was a positive result in a participant who was diagnosed with breast cancer by further diagnostic work-up. A false-positive screening result was a positive result in the absence of breast cancer. A true-negative screening result (specificity) was a negative result in the absence of breast cancer and a false-negative test result was a negative result followed by diagnosis of interval cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zheng, Study Chair — Fudan University
Locations (3):
- China (3):
  - Maternal and Infant Healthy Centre of Hongkou District, Shanghai, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pudong New Area Healthcare Hospital For Women & Children, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results. And the data will only be transferred after signing of a data access agreement.
Access Criteria: The study chairman will consider access to study data upon written detailed request sent to her, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Shen J, Liu Y, Liu A, Gu X, Zhou J, Jiang P, Mo M, Zhang L, Yang C, Zhou C, Wang Z, Xie Z, Yao W, Zhou S, Zheng Y, Chang C. Artificial intelligence-assisted ultrasound screening for breast cancer in China: a prospective, clustered, controlled, population-based study. Breast Cancer Res. 2025 Oct 7;27(1):173. doi: 10.1186/s13058-025-02128-0. PMID 41057952

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT06521788/Prot_SAP_000.pdf